CLINICAL TRIAL: NCT03871582
Title: Number of Meals With Adequate Protein Intake and Functionality in Middle to Older Aged Mexican Adults
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Hospital General de Occidente (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Sport, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: HGO-ICAAFYD18-3
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Aging
Keywords: Protein intake; Older adults; Mexican adults; Functionality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Middle to older aged (>50 years) Mexican adults attending to the Geriatrics Department from the Western General Hospital (Zapopan, Jalisco,Mexico).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
The objective of this study was to analyze if the number of meals with adequate protein intake is associated with functionality in middle to older aged mexican adults.

DETAILED DESCRIPTION:
Dietary protein intake per meal was assessed with 24-h dietary recalls to determine the number of meals with adequate protein intake (>30 g, >0.4 g/kg). Functionality was assessed with self-reported questionnaires about daily living activities (Barthel), and instrumental activities of daily living (Lawton). Subjects were categorized according the number of meals with adequate protein intake (zero meals, one meal, two or three meals), and their functionality score for both questionnaires (high, middle, and low scores).

With multinomial logistic regression, the investigators assessed if consuming zero or one meal with adequate protein intake could be associated with lower functionality in comparison with consuming two or three meals with enough protein. The logistic regression was adjusted for covariables (age, sex, BMI categories for the elderly, number of diagnosed diseases, inadequate protein intake per day [<1.2 g/kg/d]).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to stand up and walk independently or with walking sticks only.
* Subjects able to answer questionnaires independently or with minimum caregivers' assistance

Exclusion Criteria:

* Subjects reporting any kind of hospitalization within the last year.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle to older aged Mexican adults attending to the Geriatrics Department at the Western General Hospital (Hospital General de Occidente) for their usual medical screening or first time assessment.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Functionality on Instrumental Activities of Daily Living - Lawton questionnaire | One day
  Functionality score for instrumental activities of daily living (assessed with Lawton questionnaire). This instrument assess how well the subject perform some daily activities involving tools (e.g. handling finances, taking medication, using the telephone). The instrument consists on five items for men and eight for women, and each item is coded for 0 or 1 depending on if subjects are capable to successfully complete the activity. Therefore, the score ranges from 0 to 5 in men and 0 to 8 in women, the higher the score, the more functional the subj
Functionality on Activities of Daily Living - Barthel questionnaire | One day
  Functionality score for activities of daily living (assessed with Barthel questionnaire). This instrument assess how well the subject perform some daily activities (e.g. dressing, using stairs). The instrument consists on ten items for both men and women coded as 0 or multiples of 5 (i.e. 5, 10, 15) depending on if subjects are capable to successfully complete the activity. The score ranges from 0 to 100 for both men and women, the higher the score, the more functional the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gaytán-González, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided